CLINICAL TRIAL: NCT04929899
Title: Improving Chemotherapy-induced Nausea Control Through Bright Ideas®-CIN Training: a Feasibility Study in Children Receiving Oral Chemotherapy
Brief Title: Bright Ideas - CIN Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); Inova Fairfax Hospital (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Lee Dupuis, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000073003
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bright Ideas- CIN Training (Other): The PSST will be delivered by a "trainer" in a minimum of three 30-minute to 1-hour sessions with a parent and patient (if developmentally appropriate).
  During the first session, the study team member will build rapport by understanding relevant personal background and medical information; introduce PSST and the Bright IDEAS paradigm; review the patients experience with nausea as reported in Phase 1 and at other times during treatment; promote problem-solving strategies and skills; and develop an anti-nausea action plan. During the second session, the trainer will discuss how well the prior action plan worked and reinforce successful outcomes or, if unsuccessful, return to the problem-solving steps to generate a new action plan. The third session will review progress on CINV control, assist in problem-solving as needed, and discuss how to continue to use the Bright IDEAS framework to resolve future issues with CINV or symptom management more broadly.
  Interventions: Behavioral: Bright Ideas - CIN Training

INTERVENTIONS:
Behavioral: Bright Ideas - CIN Training — Bright IDEAS is a validated problem-solving skill training intervention.

SUMMARY:
In this study investigators will determine the feasibility of a future trial comparing chemotherapy-induced nausea control in children with ALL receiving oral 6-mercaptopurine who do and do not receive problem-solving skill training. This is a novel approach to controlling an important and common treatment-related symptom.

DETAILED DESCRIPTION:
This study will evaluate a novel approach to controlling a treatment-related symptom that detracts significantly from the quality of life of many patients. It will preserve and enhance the patient's and family's autonomy with respect to self-care. If found to be effective, this approach may be generalizable to pediatric patients receiving chemotherapy other than 6-mercaptopurine and thus has the potential to improve the quality of life of many children receiving cancer therapy.

This study will evaluate the efficacy of Bright IDEAS-CIN, adapted from the validated Bright IDEAS framework to improve CIN control in children with ALL who experience nausea while receiving 6-mercaptopurine. Bright IDEAS is an 8-session face-to-face intervention with a caregiver. In this first session, the caregiver is taught the problem-solving framework and begins working on their first self-selected problem. Sessions 2-7 involve working through relevant problems, with most caregivers working through 3-4 different problems. The final session summarizes the skills and discusses how to continue to use these new skills for new problems instead of lapsing into old ineffective strategies. Investigators adapted Bright IDEAS to meet the specific problem of CINV by adapting it to 3 sessions focused specifically on CINV, including the child in the conversation when developmentally appropriate and allowing the latter sessions to be conducted by phone or video-chat.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 4 years (PeNAT validated in patients 4 to 18 yrs)
* newly diagnosed or recurrent disease: first diagnosis of ALL (i.e. non-relapsed) in maintenance therapy
* English, French or Spanish-speaking with an English, French or Spanish-speaking guardian (PeNAT available in these languages)
* without physical or cognitive impairments that preclude use of the PeNAT
* planned to receive PO 6-mercaptopurine
* not planned to receive IV, IM, SC or IT chemotherapy or oral or IV corticosteroids during the 7-day study period

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percent of eligible patients who consent/assent to participate and completion of study procedures by 20 patients within 24 months | 24 months from study activation
  A future trial will be feasible if
  * 50% of patients deemed to be eligible to participate in Phase 1 consent/assent to participate
  * the recruitment into Phase 2 of 20 evaluable patients across all participating centers within 24 months of study activation of whom 80% return a completed CINV diary for at least 5 days of each 7-day data collection period. A completed CINV diary contains at least one PeNAT score and a record of the time of each vomiting episode or noting the presence/absence of vomiting daily. Evaluable patients are defined as those who have completed at least one cycle of PSST.

SECONDARY OUTCOMES:
CIN and CIV incidence | 24 months from study activation
  Proportion of children who report CIN and chemotherapy-induced vomiting (CIV) in Phase 1 and Phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dupuis, PhD, Principal Investigator — SickKids Research Institute
Locations (4):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Inova Children's Hospital, Falls Church, Virginia
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No